CLINICAL TRIAL: NCT05457309
Title: Construction and Effect Evaluation of Malignant Fungating Wounds Care Regimen for Breast Cancer Patients Based on Symptom Management Theory
Brief Title: Construction and Effect Evaluation of Malignant Fungating Wounds Care Regimen for Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-024-01
Record Dates: First submitted 2022-06-24; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Malignant Fungating Wound
Keywords: Breast cancer; Malignant fungating wounds; Symptom management; Wound care; Quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- malignant fungating wounds care regimen (Experimental): malignant fungating wounds care regimen based on the evidences, expert consultation, pre-experiment and final determination
  Interventions: Procedure: malignant fungating wounds care regimen

INTERVENTIONS:
Procedure: malignant fungating wounds care regimen — 1) Preliminary construction of regimen: The researchers summarized the literatures and guidelines about malignant fungating wounds care, and then formed a preliminary draft of the regimen.2) Expert consultation: Experts in malignant fungating wound care, breast cancer and rehabilitation were consulted by email, and the researchers revised the protocol according to the experts' comments, and the final draft was determined after multiple rounds of consultation with experts. 3) Pre-experiment: The researchers investigated the enrolled patients to assess the feasibility of the protocol, and adjusted the content based on the feedback.4) Final Determining: including health records establishment, the intervention time, implementers, location, method and frequency. A wound care team was formed, interventions were carried out in terms of somatic care, wound home care, psychological support, and rehabilitation guidance, and the enrolled patients would be regularly followed by the researchers.

SUMMARY:
Patients with breast cancer malignant fungating wounds have six specific symptoms caused by wounds: malodor, pain, massive exudate, bleeding, infection, and pruritus. Malignant fungating wounds cause patients' physical condition and social function to be severely restricted, and the cost of wound dressing change further increases financial pressure, which leads to low self-identity, complex and variable emotions, and low quality of life. Therefore, the care of patients with malignant fungating wounds focuses on symptom management with the aim of improving the quality of life. There are scarce well-defined wound symptom management programs for this group, and most focus on wound management while ignoring the impact on the patient's body and mind. This study will construct malignant fungating wounds care regimen for breast cancer patients in order to improve the quality of life.

DETAILED DESCRIPTION:
Patients with breast cancer malignant fungating wounds have six specific symptoms caused by wounds: malodor, pain, massive exudate, bleeding, infection, and pruritus, and there is an interrelationship between the symptoms. The symptoms presented by patients have certain individual differences and vary with the stage of treatment and treatment effect, which bring different degrees of distress to patients and their families and seriously affect patients' prognosis and quality of life. It is found that wound symptoms such as malodor are significantly negatively correlated with the quality of life of patients with malignant fungating wounds. Malignant fungating wounds cause patients' physical condition and social function to be severely restricted, and the cost of wound dressing change further increases financial pressure, which leads to low self-identity, complex and variable emotions, and low quality of life. With the continuous improvement of cancer treatment level, patients' quality of life is more representative of cure and recovery than survival to some extent. Therefore, the care of patients with malignant fungating wounds focuses on symptom management with the aim of improving the quality of life. There are scarce well-defined wound symptom management programs for this group, and most focus on wound management while ignoring the impact on the patient's body and mind. This study will take the symptom management theory as the guide, start from the actual needs of patients and combine with the actual clinical situation to construct malignant fungating wounds care regimen for breast cancer patients in order to improve the quality of life and make their lives dignified and meaningful.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old with pathologically confirmed diagnosis of breast cancer.

  * Tumor metastasis in the chest wall or other sites and rupture to form a malignant fungating wound with a wound area of at least 10cm2 or more.

    * Knowing of the cancer diagnosis. ④ Capable and willing to receive follow-up.

      * Informed consent and voluntary participation.

Exclusion Criteria:

* Patients with mental illness or cognitive impairment and language expression deficiency.

  * Patients with extensive metastasis of cancer throughout the body to the chest, shoulders, back, arms, etc. and whose treatment was ineffective.

    * Patients at the end stage of death.

      * Patients who refused to participate in this study.

Withdrawal criteria:

* Patients who developed serious complications during the study and were unable to continue the study.

  * Patients who died during the study. ③Patients who requested withdrawal on their own during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-06-24 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Wound Size at day 42 | Baseline and day 42
  described by "healing, improvement, maintenance, deterioration", where "wound healing" refers to 100% epithelialization of the wound, "wound improvement" refers to reduction of the wound area, "wound maintenance" refers to no change in the wound area, and "wound deterioration" refers to an increase in the wound area.

SECONDARY OUTCOMES:
Change from Baseline in Wound symptoms at day 42 | Baseline and day 42
  measured using the scale named "Toronto Symptom Assessment System for Wound(TSAS-W)"; the minimum and maximum values are 0 and 100 respectively, and higher scores mean a worse wound symptom reported by patients.
Change from Baseline in Quality of life in breast cancer patients at day 42 | Baseline and day 42
  measured using the scale named "Quality of Life instruments for Cancer Patients-Breast Cancer(QLICP-BR)". There are 37 items, and 5~10 and 27~32 are positive entries, and the rest are reverse entries. Using Likert 5-level scoring method, the total score is 36~180 points. The higher the total score, the better the quality of life. Only 35 items were used in this study.
Change from Baseline in Social support at day 42 | Baseline and day 42
  measured using the scale named "Social Support Rate Scale(SSRS)".The scale includes 10 items and 3 dimensions, with a total score of 11-59. The higher the total score, the better the social support.
Change from Baseline in Anxiety at day 42 | Baseline and day 42
  measured using the scale named "Self-rating Anxiety Scale(SAS)". SAS scale includes 20 items. If it is a positive scoring question, it will be rated as rough score 1, 2, 3 and 4 in turn; Reverse scoring questions (those with * sign) will be rated as 4, 3, 2, 1 points. Add the scores of 20 items to get the rough score (x). Multiply the rough score by 1.25 and take the integer part to get the standard score (y). According to the results of the Chinese norm, the cut-off value of SAS standard deviation is 50 points, of which 50 ~ 59 points are mild anxiety, 60 ~ 69 points are moderate anxiety, and more than 70 points are severe anxiety.
Change from Baseline in Depression at day 42 | Baseline and day 42
  measured using the scale named "Self-rating Depression Scale(SDS)". SDS scale includes 20 items and 10 positive scoring questions, which are rated as rough scores of 1, 2, 3 and 4 in turn; 10 reverse scoring questions (those with * sign) will be rated as 4, 3, 2, 1 points. Add the scores of 20 items to get the rough score (x). Multiply the rough score by 1.25 and take the integer part to get the standard score (y). According to the results of the Chinese norm, the cut-off value of SDS standard score is 53 points, of which 53-62 points are mild depression, 63-72 points are moderate depression, and more than 73 points are severe depression.
Change from Baseline in Stigma at day 42 | Baseline and day 42
  measured using the scale named "Stigma Scale for Chronic Illness 8-item version(SSCI-8items)". The scale is developed on the basis of the 24 item stigma scale for chronic illness (SSCI), with a total of 8 items, of which 3 items are from internal shame, 5 items are from external shame, and all items are positive. The five options of the scale are: No, little, sometimes, often, always, and assigned 1, 2, 3, 4, and 5 points respectively, with a total score of 8 to 40 points. The higher the score, the higher the level of shame.

OTHER OUTCOMES:
Change from Baseline in Wound bleeding at day 42 | Baseline and day 42
  Patients were counted to self-report the number and severity of wound bleeding in the recent 1-week period, the severity of wound bleeding was reported by the patient using a scale of 1~10, and higher scores mean a more severe and frequent wound bleeding reported by patients in the last week.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen memorial hospital, Sun Yat-sen university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No